CLINICAL TRIAL: NCT00673803
Title: Influence of Two Sharp-edged Hydrophobic Acrylic Micro-incision-IOLs on Posterior Capsule Opacification. A Randomized, Double-masked Study With Intraindividual Comparison.
Brief Title: Influence of Two Different Preloaded Intraocular Lens (IOLs) on Posterior Capsule Opacification
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Hietzing (Other)
Responsible Party: Matthias Wirtitsch MD, Hietzing Hospital, Vienna, Austria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: preloaded 2008
Record Dates: First submitted 2008-05-06; First posted 2008-05-07 (Estimated); Last update posted 2010-08-17 (Estimated); Status verified 2008-12

CONDITIONS: Cataract
Keywords: posterior capsule opacification; micro incision; sharp optic edge
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Other): cataract surgery, implantation of a Polylens Y10
  Interventions: Procedure: cataract surgery
- B (Other): cataract surgery, implantation of a Polylens Y30
  Interventions: Procedure: cataract surgery

INTERVENTIONS:
Procedure: cataract surgery — cataract surgery with implantation of an IOL
  Other Names: Polylens Y30 IOL, Polytech, Germany; Polylens Y10 IOL, Polytech, Germany

SUMMARY:
Studies showed that a sharp posterior optic edge of an intraocular lens (IOL) inhibits migration of lens epithelial cells in between posterior capsule and optic of the IOL and therefore reduces the rate of posterior capsule opacification (PCO). In present time most IOLs implanted have a sharp posterior optic edge. Due to differences in IOL production different IOLs have different rates of PCO.

Progression in cataract surgery technique allow phacoemulsification through micro-incisions. Therefore there is need for IOLs that can be implanted through incisions of about 2.5 mm.

This study investigates the effect of two different hydrophobic acrylic IOLs with a sharp posterior optic edge on the rate of PCO after implantation through a micro-incision. The results will be compared intraindividually.

DETAILED DESCRIPTION:
prospective, randomized, bilateral study with intraindividual comparison, implantation of a Polylens Y10 IOL in one eye and implantation of a Polylens Y30 in the contralateral eye.

PCO rate will be detected at 1 year and 2 years.

ELIGIBILITY:
Inclusion Criteria:

* bilateral age-related cataract
* age 55 to 80 years
* expected postoperative visual acuity of at least 0.5

Exclusion Criteria:

* amblyopia
* corneal scars
* diabetes
* pseudoexfoliation-syndrome
* earlier ocular surgeries or laser treatments
* intraocular tumors

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-12; Primary Completion 2009-07 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
PCO rate | 2 years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Nadja Karnik, MD, Study Chair — Dept of Ophthalmology, Hietzing Hospital, Vienna, Austria
Locations (1):
- Department of Ophthalmology, Hietzing Hospital, Vienna, Austria